CLINICAL TRIAL: NCT04736004
Title: Hearts of Athletes Study: Prospective Evaluation of Athletes for Cardiac Involvement With COVID-19
Brief Title: Hearts of Athletes
Status: Terminated | Type: Observational
Why Stopped: Study terminated due to insufficient participant enrollment during the COVID-19 pandemic, which impacted recruitment timelines and feasibility of meeting study objectives.
Sponsor: Duke University (Other)
Collaborators: The Joel Cornette Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: Pro00106943
Record Dates: First submitted 2021-01-29; First posted 2021-02-03 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Cardiac Involvement With COVID-19
Keywords: athletes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Athletes with COVID-19
- Athletes without COVID-19 (control)

SUMMARY:
The Hearts of Athletes study is being conducted to determine the heart involvement with COVID-19 in athletes. This study aims to enroll any Adult (18 years of age or greater)

• Athlete is defined as NCAA Collegiate Athlete, Professional Athlete, Military, or Olympic Athlete will be eligible for the study.

With COVID-19

• COVID-19 diagnosed via an RT-PCR (nasal or throat swab test) prior to enrollment

Or without COVID-19

• Identified as a local Control participant (similar sport) to a participant with COVID-19, who is willing to undergo a standard cardiovascular evaluation

Participants with and without COVID-19 will use their mobile devices to provide health information, like symptoms, by answering survey questions daily for 30 days. Also, participants will allow their de-identified cardiac images to be sent to the Duke Heart Center for blinded analysis.

No physical risks are associated with this study. One possible risk, although minimal, is loss of confidentiality.

ELIGIBILITY:
Inclusion Criteria:

* Any adult athlete (defined as NCAA Collegiate Athlete, Professional Athlete, or Olympic Athlete) will be eligible for the study.
* COVID-19 diagnosed via an RT-PCR, or history of COVID-19 antibodies at least 10 days and less than 6 months prior to consent
* No longer requiring quarantine per local health recommendations, prior to cardiovascular evaluation.
* Identification as a Control participant (similar sport) to a participant without COVID-19 willing to undergo cardiovascular evaluation

Exclusion Criteria:

* Anyone with known cardiovascular disease - defined as known myocardial disease, valvular heart disease, or known coronary heart disease
* Anyone without the ability to provide informed consent
* Anyone with a known contraindication to cardiac magnetic resonance (metallic implant)

Ages: 18 Years to 30 Years | Sex: All
Age Groups: Adult
Study Population: Any adult athlete, defined as NCAA Collegiate Athlete, Professional Athlete, or Olympic Athlete, with COVID-19 compared to any adult athlete without COVID-19.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2022-11-03 (Actual); Primary Completion 2025-09-24 (Actual); Study Completion 2025-09-24 (Actual)

PRIMARY OUTCOMES:
Rate of Definite Myocarditis as measured by CMR (Cardiac Magnetic Resonance Imaging) | Up to 7 months
Rate of Possible Myocarditis as measured by CMR (Cardiac Magnetic Resonance Imaging) | Up to 7 months

SECONDARY OUTCOMES:
Number of abnormal ECGs as measured by medical record abstraction | Up to 7 months
Number of abnormal Troponin as measured by medical record abstraction | Up to 7 months
Number of abnormal echocardiogram as measured by medical record abstraction | Up to 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Manesh Patel, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No